CLINICAL TRIAL: NCT06162923
Title: The Effectiveness of Reinforcement of Oral Hygiene Education Through Video During Fixed Orthodontic Treatment in Adults -A Randomised Clinical Trial
Brief Title: The Effectiveness of Reinforcement of Oral Hygiene Education Through Video During Fixed Orthodontic Treatment in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DrOrtho LPL
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Oral Hygiene Reinforcement During Fixed Orthodontic Treatment
Keywords: Oral hygiene reinforcement; video; fixed orthodontic treatment; adult

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to three groups (control group, onsite video group and remote video group) at a 1:1:1 ratio in this three-arm parallel.
Who Masked: Investigator, Outcomes Assessor
Masking Description: This is a randomised, single-blind clinical trial. Because the allocation sequence and types of interventions delivered to the participants will be performed by an independent clinician, the main investigator can be blinded to the types of interventions that the participants will receive. The main clinician will be in charge of data collection. The data will be passed to the independent clinician once the main clinician has completed data collection. The data will be entered into the Data Collection Sheet by the independent clinician, who will also generate coding for the participants' names and types of interventions. The data is then passed to the main clinician for analysis. As a result, the main clinician is also blinded during the data analysis stage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention)
- On-site video group (Experimental)
  Interventions: Behavioral: On-site video group
- Remote video group (Experimental)
  Interventions: Behavioral: Remote video group

INTERVENTIONS:
Behavioral: On-site video group — Each participant will receive standard oral hygiene reinforcement verbally, followed by watching a pre-recorded oral hygiene instruction video on a tablet
  Arms: On-site video group
Behavioral: Remote video group — After receiving normal oral hygiene reinforcement verbally, each participant will be sent a video link Whatapps instant message, which they are required to watch at home
  Arms: Remote video group

SUMMARY:
Effective oral hygiene education is paramount to ensure lasting good oral hygiene habits in patients receiving fixed orthodontic treatment. Repetition and reinforcement play an important role in the sustainability of oral health behaviour. Video-based oral hygiene education can be provided in chairside, or it can be provided to the participant to watch at home, saving clinicians a lot of time. The study aims to investigate the long-term effects of different methods of video-assisted oral hygiene reinforcement on the oral hygiene of participants receiving fixed orthodontic treatment, as well as the consequences when reinforcement is discontinued. Sixty participants will be randomly allocated to three groups at a 1:1:1 ratio in this three-arm parallel, randomized clinical trial. Sixty participants will be randomly allocated to the control group, study group 1 (onsite video) and study group 2 (remote video). The Orthodontic Plaque Index (OPI) and Full-mouth Bleeding Score (FMBS) will be measured at baseline and every two months for up to 12 months. Following data collection, statistical data analysis will be conducted to compare the outcomes and changes between the three groups.

DETAILED DESCRIPTION:
Orthodontic treatment is a technique for straightening teeth or correcting malocclusions that has many recognised benefits, including improved aesthetics and patient self-esteem. Rapid advances in orthodontic treatment have broadened the area of treatment to include not just children and adolescents, but even adults. Adult patients seeking orthodontic treatment have increased in number over the past few years, for a variety of reasons, the most prevalent of which is the desire to straighten their teeth and improve their smile.

The key to successful orthodontic treatment is correcting occlusion in the best feasible way to improve aesthetics and function while preserving the pre-existing health of teeth and supporting tissues. Fixed appliances increase the retention areas for plaque accumulation, and this often makes maintaining optimal self-performed oral hygiene a challenge for the patients. Dental plaque that builds upon the orthodontic brackets in a poor oral environment consists of pathogenic biofilms that can lead to undesirable complications such as white spot lesions, gingivitis, and periodontal breakdown. Moreover, poor oral hygiene during orthodontic treatment often results in poor treatment quality and prolonged treatment duration. Poor oral hygiene is estimated to be the reason for 5%-10% of orthodontic patients failing to complete treatment.

Successful orthodontic treatment requires the patient's cooperation, in particular the maintenance of oral hygiene, which is controlled by the patient throughout the orthodontic treatment. Studies have indicated that minimal periodontal disease, bone loss, and cavities will occur throughout the course of fixed orthodontic treatment provided proper plaque control measures are implemented. In order to achieve optimal oral hygiene, professionals must provide detailed and understandable instructions, as well as suitable equipment and patient motivation, which is crucial for ensuring compliance. However, adequate plaque control still necessitates that each individual engages in regular oral hygiene behaviours. It is difficult to ensure patient compliance with home care recommendations, and as a result, long-term treatments such as orthodontic frequently have only a 50% compliance rate.

In dentistry, education is utilised to increase patient knowledge growth since it has the greatest influence on behavioural change, particularly with regard to oral hygiene. It has been demonstrated that repetition and reinforcement play an important role in the sustainability of health behaviour. Previous studies of oral health education have found that oral health educational programmes can only provide short-term improvements in oral health behaviour and oral health status, and this is especially true for most of the single session programs. Furthermore, Cozzani, in his study, found that post-procedural communication between the orthodontist and patient is an important element in improving dental hygiene compliance. By fostering mutual trust, the orthodontist may ensure that oral hygiene instructions are followed more consistently and educate patients about the benefits of behaving properly. Therefore, oral health education should be a continuous effort, and repetition and reinforcement are crucial to the long-term success of oral health educational programmes. As fixed orthodontic treatment can take more than two years to complete and requires patient compliance with perfect oral hygiene throughout the treatment, repetition and reinforcement of oral hygiene education play a significant role in the sustainability of good oral hygiene behaviour.

In dentistry, many studies have been conducted to assess the effectiveness of various oral health educational strategies in encouraging behavioural changes in patients undergoing fixed appliance orthodontic treatment. A variety of techniques, including verbal communication, written material with pictures, videos, and visual demonstration using models or experimental tools like indicator dyes or displaying live bacteria to patients under a phase contrast microscope, have been used. Although the one-to-one approach to oral health education is promising in terms of improving oral hygiene, it is time-consuming and impractical. With technological advancements and increased internet availability, the use of videos as electronic health education material is gaining acceptability and becoming an appealing medium for communicating information to patients. Video-based oral hygiene education can be presented in a variety of methods, such as chairside, where patients are required to watch the video in the clinic, or it can be provided to the patient to watch at home.

To the best of the investigators knowledge, no study has been done to assess the influence of different methods of video-assisted oral hygiene reinforcement in improving patients' oral hygiene throughout fixed orthodontic treatment and minimal studies on the impacts of oral hygiene reinforcement have been undertaken purely on adult patients. Based on the available data, the majority of the studies did not look into the outcomes for the patients' oral health in more detail after discontinuing the oral hygiene reinforcement. Therefore, the impacts of oral hygiene reinforcement via different video delivery methods will give crucial data and insight into the oral health outcomes of adult patients receiving fixed orthodontic treatment, and we would also like to study the effects when the oral hygiene reinforcement is discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Require fixed orthodontic treatment in upper and lower arches
* Agree to use conventional stainless-steel brackets
* Full-Mouth Plaque Score of 40-70%
* Absence of caries and overhanging or distorted restoration
* Stable or no periodontal diseases with the presence of Basic Periodontal Examination (BPE) code 0/1/2 with no obvious evidence of interdental recession
* Have at least 20 teeth (Ozlu et al., 2021)
* Capable of using and accessing technology gadgets such as a smartphone, tablet, laptop, and computer
* Having access to the internet and having WhatsApp's account

Exclusion Criteria:

* Presence of BPE code 3/4
* Presence of current active periodontal disease
* Smokers
* Severe or chronic illnesses (such as diabetes, cardiovascular diseases, stroke, etc)
* Physically impaired and syndromic patient
* Orofacial deformities
* History of previous orthodontic treatment
* Intake of antibiotics within 6 months before and during the study period
* Taking drugs that influence gingival inflammation or bleeding (eg anticoagulants, cortisone)
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Orthodontic Plaque Index (OPI) | Every two months for up to 12 months
  The plaque deposits around the brackets will be disclosed using a disclosing solution to facilitate their detection. The dentition is divided into six sextants. The amount of plaque accumulation on each tooth surface at the bracket base (mesial, distal, occlusal/incisal, and cervical) is represented by a score ranging from 0 to 4. 0 represents best outcome whereas 4 represents worst outcome.

SECONDARY OUTCOMES:
Full-Mouth Bleeding Score (FMBS) | Every two months for up to 12 months
  Presence or absence of gingival bleeding on each tooth surface (mesial, distal, buccal and lingual/palatal) in the dentition is recorded in a dichotomous manner. The FMBS will be performed through gentle probing of the gingival crevice on each tooth surface. A positive finding will be recorded if bleeding occurs within 10 seconds. Yes represents the presence of bleeding (worse outcome) and no represents the absence of bleeding (better outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Universiti Malaya, Kuala Lumpur, Malaysia